CLINICAL TRIAL: NCT04615286
Title: Short Versus Long Antibiotic Course for Pleural Infection Management (SLIM Trial): a Randomized Controlled Open Label Trial
Brief Title: Short Versus Long Antibiotic Course for Pleural Infection Management (SLIM Trial)
Acronym: SLIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3/24/11/10/2020
Record Dates: First submitted 2020-10-14; First posted 2020-11-04 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Pleural Infection
MeSH Terms: interventions — Anti-Bacterial Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short course (Experimental): Antibiotic course of 2-3 weeks overall duration for treating pleural infection
  Interventions: Other: Short course (2-3 weeks) of antibiotics
- Long course (Active Comparator): Antibiotic course of 4-6 weeks overall duration for treating pleural infection
  Interventions: Other: Standard (long course) of antibiotics

INTERVENTIONS:
Other: Short course (2-3 weeks) of antibiotics — Shorter course of antibiotic than standard care of 4-6 weeks
  Arms: Short course
Other: Standard (long course) of antibiotics — 4-6 weeks of antibiotics
  Arms: Long course

SUMMARY:
Infection of the pleural space is serious condition that requires hospitalization, invasive interventions and long courses of antibiotics[1]. Treatment of pleural infection requires long hospital admission with a median of 19 days[2] and medical treatments fails requiring surgical intervention in up to 30% of cases[3]. The mortality from pleural infection is around 10% at 3 months[4].

Besides drainage of the infected fluid, antibiotics are a core component of management of pleural infection[5] and are typically given intravenously in the first few days of treatment until the condition is stabilized at which stage patients are shifted to oral antibiotics of equivalent spectrum. In almost half of the cases of pleural infection, the choice of antibiotics is entirely empirical due to low yield of microbiological tests on pleural fluid in these cases[6]. International guidelines cite a minimum length of antibiotic course of pleural infection of four weeks[5,7] with antibiotic courses typically lasting six weeks[8]. However, these recommendations are based on expert opinion with no robust evidence to support such durations.

The RAPID (renal function, age, purulence, infection source and dietary factors) score has recently been validated as a robust tool to predict 3-month mortality of patients with pleural infection based on demographic and laboratory data (table 1)[4]. A low score (0-2) is associated with 2-3% mortality, medium score (3-4) 9% mortality and high score (5-7) 30% mortality at three months[9]. The utility for this score in clinical management is yet to be determined and this study will attempt using this score to stratify lengths of antibiotic treatment based on proposed risk of adverse outcomes as stipulated by the RAPID score.

The aim of this study is to investigate the feasibility and safety of prescribing shorter courses of antibiotics (2-3 weeks) versus the standard longer courses (4-6 weeks) in medically-treated patients with pleural infection at lower risk of mortality (RAPID score 0-4) who can be safely discharged home within 14 days of hospitalization and how this impacts success of medical treatment.

DETAILED DESCRIPTION:
Infection of the pleural space is serious condition that requires hospitalization, invasive interventions and long courses of antibiotics. Treatment of pleural infection requires long hospital admission with a median of 19 days and medical treatments fails requiring surgical intervention in up to 30% of cases. The mortality from pleural infection is around 10% at 3 months.

Besides drainage of the infected fluid, antibiotics are a core component of management of pleural infection and are typically given intravenously in the first few days of treatment until the condition is stabilized at which stage patients are shifted to oral antibiotics of equivalent spectrum. In almost half of the cases of pleural infection, the choice of antibiotics is entirely empirical due to low yield of microbiological tests on pleural fluid in these cases. International guidelines cite a minimum length of antibiotic course of pleural infection of four weeks with antibiotic courses typically lasting six weeks[8]. However, these recommendations are based on expert opinion with no robust evidence to support such durations. A recent trial compared a two-week versus a three-week antibiotic course for parapneumonic pleural infections. The trial that concluded prematurely due to inability to recruit to target sample size and found that the two regimens were equivalent in terms of risk of failure of medical treatment. Besides being an underpowered study, the results are only applicable to parapneumonic effusions but not primary pleural infections.

The RAPID score has recently been validated as a robust tool to predict 3-month mortality of patients with pleural infection based on demographic and laboratory data. A low score (0-2) is associated with 2-3% mortality, medium score (3-4) 9% mortality and high score (5-7) 30% mortality at three months. The utility for this score in clinical management is yet to be determined and this study will attempt using this score to stratify lengths of antibiotic treatment based on proposed risk of adverse outcomes as stipulated by the RAPID score. A shorter antibiotic course that is as effective as the standard long course is desirable given the common occurrence of side effects with antibiotic treatment. The presence of a robust predictive score of outcome seems as an attractive tool to help stratify patients who can be safely treated with shorter antibiotic courses.

The aim of this study is to investigate the feasibility and safety of prescribing shorter courses of antibiotics (2-3 weeks) versus the standard longer courses (4-6 weeks) in medically-treated patients with pleural infection at lower risk of mortality (RAPID score 0-4) who can be safely discharged home within 14 days of hospitalization and how this impacts success of medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years old)
* Willing to provide informed consent
* Admitted to hospital for treatment of pleural infection (both parapneumonic and primary pleural infections included). Pleural infection will be defined by the presence of one of the following:

  1. the presence of pus in the pleural space;
  2. positive pleural fluid gram stain or culture; or
  3. pleural fluid pH < 7.2 or pleural fluid glucose < 40 mg/dL in the setting of acute respiratory infection.
* RAPID low or intermediate score (0-4)
* Fit for discharge within 14th day of admission

Exclusion Criteria:

* Failure of medical treatment within 14 days of admission and need for surgical referral
* Need for hospital admission beyond 14 days due to medical reasons
* Admission to recurrent ipsilateral pleural infection within the last three months
* RAPID high score (5 or more)
* Pleural infection not amenable to drainage at time of diagnosis and therefore upfront decision to treat with prolonged antibiotics
* Residual pleural collection (despite attempted drainage) that the managing clinician indicated is for prolonged oral suppressive therapy (i.e. six weeks of oral antibiotics).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2021-11-10 (Actual); Study Completion 2021-12-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with failure of medical treatment | Outcome assessed at six weeks post diagnosis
  Incidence of failure of treatment as judged by trial clinician requiring further antibiotics and/or tube drainage and/or surgical intervention by six weeks post initial admission. Failure will be determined based on the one or more of the following parameter: clinical (recurrence of symptoms), biochemical (worsening of WCC [by 2000/mm3] or CRP [by > 20%] from discharge values) and radiological (chest X-ray +/- TUS evidence of increasing or new pleural collection).

SECONDARY OUTCOMES:
Length of antibiotic treatment in days | Outcome assessed at six weeks post diagnosis
  Total length of antibiotic treatment (in days) in the study arms
Number of participants with chest X ray worsening at 6 weeks | Outcome assessed at six weeks post diagnosis
  Number of participants with worsening in the 6-week chest X-ray as compared to discharge chest X-ray in the study arms. Chest X-ray pairs (discharge vs 6-week) will be read by a respiratory physician blinded to treatment allocation who will judge whether there is worsening (versus stability or improvement)
Time to return to normal daily activities in days | Outcome assessed at six weeks post diagnosis
  Time (in days) to return to normal daily activities in participants of the study arms
Number of participants requiring readmission within 30 days from discharge | 30 days from discharge
  Readmission within 30 days from discharge

CONTACTS AND LOCATIONS:
Overall Officials: Maged Hassan, PhD, Principal Investigator — Alexandria University Faculty of Medicine
Locations (1):
- Alexandria University Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The spreadsheets with de-identified patient information will be stored securely after trial conclusion with the principal investigator and will be accessible to other members of the study team. Request to access study data by persons outside the study teams will be expected via email and access will be granted by the principal investigator if the request is deemed reasonable.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 5 years after study completion
Access Criteria: The data that support the findings of this study will be available on request from the corresponding author upon publishing the manuscript with the main results.

REFERENCES:
- [Background] Davies HE, Davies RJ, Davies CW; BTS Pleural Disease Guideline Group. Management of pleural infection in adults: British Thoracic Society Pleural Disease Guideline 2010. Thorax. 2010 Aug;65 Suppl 2:ii41-53. doi: 10.1136/thx.2010.137000. No abstract available. PMID 20696693
- [Background] Cargill TN, Hassan M, Corcoran JP, Harriss E, Asciak R, Mercer RM, McCracken DJ, Bedawi EO, Rahman NM. A systematic review of comorbidities and outcomes of adult patients with pleural infection. Eur Respir J. 2019 Oct 1;54(3):1900541. doi: 10.1183/13993003.00541-2019. Print 2019 Sep. PMID 31391221
- [Background] Maskell NA, Lee YC, Gleeson FV, Hedley EL, Pengelly G, Davies RJ. Randomized trials describing lung inflammation after pleurodesis with talc of varying particle size. Am J Respir Crit Care Med. 2004 Aug 15;170(4):377-82. doi: 10.1164/rccm.200311-1579OC. Epub 2004 May 13. PMID 15142871
- [Background] Corcoran JP, Psallidas I, Gerry S, Piccolo F, Koegelenberg CF, Saba T, Daneshvar C, Fairbairn I, Heinink R, West A, Stanton AE, Holme J, Kastelik JA, Steer H, Downer NJ, Haris M, Baker EH, Everett CF, Pepperell J, Bewick T, Yarmus L, Maldonado F, Khan B, Hart-Thomas A, Hands G, Warwick G, De Fonseka D, Hassan M, Munavvar M, Guhan A, Shahidi M, Pogson Z, Dowson L, Popowicz ND, Saba J, Ward NR, Hallifax RJ, Dobson M, Shaw R, Hedley EL, Sabia A, Robinson B, Collins GS, Davies HE, Yu LM, Miller RF, Maskell NA, Rahman NM. Prospective validation of the RAPID clinical risk prediction score in adult patients with pleural infection: the PILOT study. Eur Respir J. 2020 Nov 26;56(5):2000130. doi: 10.1183/13993003.00130-2020. Print 2020 Nov. PMID 32675200
- [Background] Bedawi EO, Hassan M, Rahman NM. Recent developments in the management of pleural infection: A comprehensive review. Clin Respir J. 2018 Aug;12(8):2309-2320. doi: 10.1111/crj.12941. PMID 30005142
- [Background] Hassan M, Cargill T, Harriss E, Asciak R, Mercer RM, Bedawi EO, McCracken DJ, Psallidas I, Corcoran JP, Rahman NM. The microbiology of pleural infection in adults: a systematic review. Eur Respir J. 2019 Oct 1;54(3):1900542. doi: 10.1183/13993003.00542-2019. Print 2019 Sep. PMID 31248959
- [Background] Bhatnagar R, Maskell N. The modern diagnosis and management of pleural effusions. BMJ. 2015 Sep 8;351:h4520. doi: 10.1136/bmj.h4520. No abstract available. PMID 26350935
- [Background] Hooper CE, Edey AJ, Wallis A, Clive AO, Morley A, White P, Medford AR, Harvey JE, Darby M, Zahan-Evans N, Maskell NA. Pleural irrigation trial (PIT): a randomised controlled trial of pleural irrigation with normal saline versus standard care in patients with pleural infection. Eur Respir J. 2015 Aug;46(2):456-63. doi: 10.1183/09031936.00147214. Epub 2015 May 28. PMID 26022948
- [Background] Rahman NM, Kahan BC, Miller RF, Gleeson FV, Nunn AJ, Maskell NA. A clinical score (RAPID) to identify those at risk for poor outcome at presentation in patients with pleural infection. Chest. 2014 Apr;145(4):848-855. doi: 10.1378/chest.13-1558. PMID 24264558

DOCUMENTS (1):
  • Study Protocol (2020-10-13): https://cdn.clinicaltrials.gov/large-docs/86/NCT04615286/Prot_000.pdf